CLINICAL TRIAL: NCT00196456
Title: Photodynamic Lasertherapy (PDT) in Periodontal Treatment (in Vivo)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: III UV 06/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Periodontal Disease
Keywords: Photodynamic lasertherapy; Periodontol disease
MeSH Terms: conditions — Periodontal Diseases

INTERVENTIONS:
Procedure: photosensitisation

SUMMARY:
The purpose of the study is to evaluate the effect of the photodynamic therapy in periodontal patients

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effect of the photodynamic therapy in periodontal pockets and to assess the reduction of subgingival bacteria.

The first step will include the evaluation of the quantity of the light which will activate the photosensitizer in the various niches in the periodontal pocket.

The second step will evaluate the distribution of the photosensitizer in the periodontal pocket.

The third step will assess the woundhealing of the the photodynamic therapy compared to conventional periodontal therapy with an ultrasonic device.

ELIGIBILITY:
Inclusion Criteria:

* systemic healthy
* >15 teeth
* ≤ 6 mm >2 teeth
* age > 35 years

Exclusion Criteria:

* - systemic ill
* cardiac pacemaker
* < 15 teeth

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-04; Study Completion 2005-01

PRIMARY OUTCOMES:
pocket depth reduction

SECONDARY OUTCOMES:
attachmentlevel loss

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kocher, Prof.Dr., Principal Investigator — Ernst-Moritz-Arndt University Greifswald
Locations (1):
- Ernst-Moritz-Arndt-Universität Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Komerik N, Wilson M, Poole S. The effect of photodynamic action on two virulence factors of gram-negative bacteria. Photochem Photobiol. 2000 Nov;72(5):676-80. doi: 10.1562/0031-8655(2000)0722.0.co;2. PMID 11107854